CLINICAL TRIAL: NCT01773863
Title: Major Adverse Cardiac and Cerebrovascular Events in Hospitalized Patients With Community-acquired Pneumonia
Brief Title: MACCE in Hospitalized Patients With Community-acquired Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Violi, Director, Head of Internal Medicine, Clinical Professor, University of Roma La Sapienza
Other Study IDs: MACCE and CAP
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Community-acquired Pneumonia
Keywords: Community-acquired pneumonia; Acute myocardial infarction; Platelet activation; Coagulation abnormalities,; Thrombosis; Isoprosantes; NADPH oxidase; Major adverse cardiac and cerebrovascular events
MeSH Terms: conditions — Community-Acquired Pneumonia; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and urine samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Community-acquired pneumonia is the most common infection leading to hospitalization in intensive care units and the most common cause of death associated with infection disease.

Epidemiological studies have shown that respiratory tract infections are associated with an increased risk for the development of acute cardiovascular and cerebrovascular events.

This link is further supported by studies indicating that influenza vaccination is associated with a reduced risk of hospitalization for pneumonia as well as heart disease and cerebrovascular disease.

Data connecting acute respiratory tract infections and cardiovascular events stem almost exclusively from cross-sectional or retrospective studies. Thus the real incidence and the prognostic impact of AMI, as well as the pathophysiological relationship between pneumonia and cardiovascular damage is still elusive.

Inflammation plays a major role in the pathogenesis of coronary artery disease. The increased concentrations of proinflammatory cytokines together with the activation of coagulation, the down-regulation of anticoagulant mechanisms and the enhanced platelet aggregation may trigger atheroma's instability, plaque rupture and thrombus formation.

Inflammation and coagulopathy are also considered universal host responses to infection in patients with severe sepsis. Thus far limited data are available on the changes in these high regulated systems, together with platelet activity in patients with CAP and their potential relationship with cardiovascular risk.

This project will consist in a prospective multicenter study to investigate the incidence of major adverse cardiac and cerebrovascular events (MACCE) in hospitalized patients with CAP, its prognostic relevance and the potential relationship between enhanced cardiovascular risk and the activation of inflammation, coagulation and platelet aggregation in this setting.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is the most common infection leading to hospitalization in intensive care units and the most common cause of death associated with infection disease.

Epidemiological studies have shown that respiratory tract infections are associated with an increased risk for the development of acute cardiovascular and cerebrovascular events.

This link is further supported by studies indicating that influenza vaccination is associated with a reduced risk of hospitalization for pneumonia as well as heart disease, cerebrovascular disease and the risk of death from all causes during influenza seasons in elderly.

Data connecting acute respiratory tract infections and cardiovascular events stemmed almost exclusively from cross-sectional or retrospective studies and the pathophysiological relationship between pneumonia and cardiovascular damage is still elusive.

The first aim of the study will be to analyze the prevalence of major adverse cardiac and cerebrovascular events (MACCE) in patients hospitalized for CAP, followed up for two years after hospitalization.

During hospitalization myocardial damage will be strictly monitored by measuring cardiac troponins until discharge.

Cardiac troponins are established markers of myocardial damage. Cardiac troponin elevation is seen not only in the setting of acute coronary syndromes but also in a variety of conditions not directly related to flow-limiting coronary stenosis or occlusion of the coronary arteries, such as pulmonary embolism, sepsis, heart failure and stroke. In these settings, it is well documented that elevated circulating levels of troponins are associated with poor prognosis, regardless of underlying disease.

Sparse information exists concerning the significance of troponin elevation during respiratory tract infections. Most of the studies investigated the role of troponin elevation in patients admitted in hospital for acutely exacerbated chronic obstructive pulmonary disease (COPD); only a recent study investigates specifically CAP, showing a correlation between troponin elevation and oxygenation impairment; however, the underlying mechanism was not explored.

Inflammation plays a major role in the pathogenesis of coronary artery disease. The increased concentrations of proinflammatory cytokines together with the activation of coagulation, the down-regulation of anticoagulant mechanisms and the enhanced platelet aggregation may trigger atheroma's instability, plaque rupture and thrombus formation.

Systemic coagulation abnormalities including clotting activation and inhibition of anticoagulant factors have been observed in patients with severe sepsis; in patients with CAP similar changes have been detected only in the lung compartment. Changes of clotting system activation are of potential relevance as they could elicit myocardial damage with several mechanisms including coronary ischemia and/or direct inflammation of cardiac cells. Concerning this last point it is of interest that Protein C, an anticoagulant factor with anti-inflammatory property, is reduced in severe sepsis where it correlates with disease severity and mortality. Accordingly, infusion of recombinant human activated Protein C improves survival of patients with severe sepsis due to pneumococcal pneumonia.

Until now no data exists about the behavior of Protein C in patients with CAP and its interplay with myocardial damage.

Moreover no data on platelet reactivity and activation during pneumonia exist. Very limited data is only available on common viral respiratory tract infections in which enhanced platelet reactivity has been shown.

The investigators speculated that inhibition of Protein C as well as enhanced platelet activity may be implicated in myocardial damage in patients with CAP. Therefore the investigators will perform a prospective study to investigate whether this relationship exist.

Data obtained could have important clinical consequences: new therapeutic strategies targeting these systems could prevent myocardial damage and eventually MACCEs in these patients.

ELIGIBILITY:
Inclusion Criteria:

* community-acquired pneumonia

Exclusion Criteria:

* presence of immunosuppression (HIV infection, high dose of immunosuppressive agents such as prednisone, chemotherapy);
* presence of malignancy;
* pregnancy or breast feeding;
* health care-associated pneumonia

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for community-acquired pneumonia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2011-10 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Platelet activation, clotting abnormalities, myocardial damage and inflammation in CAP patients | 2 years
  Platelet and serum thromboxane, F2-isoprostanes, NOX2-activation, serum high-sensitivity cardiac troponin T, protein C and protein S at hospital admission and at hospital discharge

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events | 2 years
  Major adverse cardiac and cerebrovascular events will be assessed during hospitalization and during the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Violi, MD, Study Chair — University of Roma La Sapienza; Roberto Cangemi, MD, Principal Investigator — University of Roma La Sapienza; Roberto Cangemi, Study Director — Sapienza - Unviersity of Rome
Locations (1):
- Internal and Medical Specialities Department - Policlinico Umberto I, Rome, Italy

REFERENCES:
- [Result] Cangemi R, Calvieri C, Bucci T, Carnevale R, Casciaro M, Rossi E, Calabrese CM, Taliani G, Grieco S, Falcone M, Palange P, Bertazzoni G, Celestini A, Pignatelli P, Violi F; SIXTUS study group. Is NOX2 upregulation implicated in myocardial injury in patients with pneumonia? Antioxid Redox Signal. 2014 Jun 20;20(18):2949-54. doi: 10.1089/ars.2013.5766. Epub 2014 Mar 14. PMID 24328853
- [Result] Cangemi R, Casciaro M, Rossi E, Calvieri C, Bucci T, Calabrese CM, Taliani G, Falcone M, Palange P, Bertazzoni G, Farcomeni A, Grieco S, Pignatelli P, Violi F; SIXTUS Study Group; SIXTUS Study Group. Platelet activation is associated with myocardial infarction in patients with pneumonia. J Am Coll Cardiol. 2014 Nov 4;64(18):1917-25. doi: 10.1016/j.jacc.2014.07.985. Epub 2014 Oct 27. PMID 25444147
- [Result] Cangemi R, Calvieri C, Falcone M, Bucci T, Bertazzoni G, Scarpellini MG, Barilla F, Taliani G, Violi F; SIXTUS Study Group. Relation of Cardiac Complications in the Early Phase of Community-Acquired Pneumonia to Long-Term Mortality and Cardiovascular Events. Am J Cardiol. 2015 Aug 15;116(4):647-51. doi: 10.1016/j.amjcard.2015.05.028. Epub 2015 May 22. PMID 26089009
- [Result] Violi F, Carnevale R, Calvieri C, Nocella C, Falcone M, Farcomeni A, Taliani G, Cangemi R; SIXTUS study group. Nox2 up-regulation is associated with an enhanced risk of atrial fibrillation in patients with pneumonia. Thorax. 2015 Oct;70(10):961-6. doi: 10.1136/thoraxjnl-2015-207178. Epub 2015 Jun 29. PMID 26123660
- [Derived] Pastori D, Menichelli D, Romiti GF, Speziale AP, Pignatelli P, Basili S, Violi F, Cangemi R. Prediction of new-onset atrial fibrillation with the C2HEST score in patients admitted with community-acquired pneumonia. Infection. 2024 Aug;52(4):1539-1546. doi: 10.1007/s15010-024-02286-x. Epub 2024 May 3. PMID 38700657
- [Derived] Cangemi R, Carnevale R, Nocella C, Calvieri C, Bartimoccia S, Frati G, Pignatelli P, Picchio V, Violi F. Low-grade endotoxemia is associated with cardiovascular events in community-acquired pneumonia. J Infect. 2024 Feb;88(2):89-94. doi: 10.1016/j.jinf.2023.11.010. Epub 2023 Nov 23. PMID 38000675